CLINICAL TRIAL: NCT02960841
Title: Effectiveness of Intracavitary Manual Lymphatic Drainage Versus Conventional Treatment in the Prevention of Perineal Trauma During Labor.
Brief Title: Effectiveness of Intracavitary Manual Lymphatic Drainage
Acronym: IMLD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidad Europea de Madrid (Other)
Responsible Party: Principal Investigator, Monica de La cueva, Principal Investigator, Universidad Europea de Madrid
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UEM_TRA_2011_01
Record Dates: First submitted 2016-11-09; First posted 2016-11-10 (Estimated); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Lymphatic Diseases
MeSH Terms: conditions — Lymphatic Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Intracavitary Manual Lymphatic Drainage (Experimental): Intracavitary Manual Lymphatic Drainage technique.
  Interventions: Other: Intracavitary Manual Lymphatic Drainage
- Conventional treatment (Active Comparator): Conventional treatment active comparator
  Interventions: Other: Conventional treatment

INTERVENTIONS:
Other: Intracavitary Manual Lymphatic Drainage
  Arms: Intracavitary Manual Lymphatic Drainage
Other: Conventional treatment
  Arms: Conventional treatment

SUMMARY:
The aim of this study was to determine the effectiveness of Intracavitary Manual Lymphatic Drainage (IMLD) in the reduction of the perineal trauma and the symptoms of vaginal edema, the prevention of complications during the expulsive and the improvement in the postpartum recovery, compared to conventional treatment during the gestation, in women with the second partum. The weekly treatment is performed from the 25th gestational week in women with vulvar edema.

ELIGIBILITY:
Inclusion Criteria:

* A sample of 49 second-trimester pregnant women with gestational edema with more than 18 years of age

Exclusion Criteria:

* Primiparous women

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2012-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Pain intensity assessed by the Visual Analogue Scale | 5 weeks